CLINICAL TRIAL: NCT03436095
Title: The Clinical Study of Bundle Measures to Improve the Success Rate of Patients With Difficult Ventilator Weaning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20173357201816
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Weaning Failure
Keywords: Bundle; difficult ventilator weaning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- research group: bundle measures to help patient to weaning ventilator
  Interventions: Other: bundle measures
- historical control group: retrospect the patients who were difficult to wean from ventilator and collect some materials to compare.
  Interventions: Other: bundle measures
- External control group: contrast other same level hospitals measures to patients who are difficult to wean ventilator.
  Interventions: Other: bundle measures

INTERVENTIONS:
Other: bundle measures — Implementation of bundle measures to improve the successful rate of weaning ventilator

SUMMARY:
Based on nutritional support, Cardiopulmonary rehabilitation and Levosimendan Bundle measures, and making beside checklist of patients with difficult ventilator weaning; Implementation of nutritional risk, respiratory function, and cardiac function assessment prior to weaning; Regulate the procedure to solve the problem of difficult-weaning patients with Non neurogenic disease in ICU. Thereby,improve the success rate of weaning patients, so as to shorten the ICU hospitalization time, reduce medical costs, reduce the complications of mechanical ventilation, improve the patient's quality of life.

DETAILED DESCRIPTION:
Older than 16 years of age, ventilator therapy more than 1 weeks, Ventilator parameters meet the standard of ventilator removal, repeated more than 3 times SBT not successful, or within a short period of time within a week of successful weaning, no other new incentives to need ventilator support again, and delayed weaning from ventilator more than 1 months.

ELIGIBILITY:
Inclusion Criteria:

Older than 16 years of age, ventilator therapy more than 1 weeks,ventilator parameters up to Weaning standard, repeated more than 3 times Spontaneous Breathing Test(SBT) not successful, or within a short period of time within a week of successful weaning, no other new incentives to re machine induced delayed more than 1 months or more offline.

-

Exclusion Criteria:

Mechanical ventilation patients who are clearly defined as neurological disorders or advanced tumor wasting diseases, as well as those without informed consent.

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: difficult-weaning patients with Non neurogenic disease in ICU.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Bundle measures can solve the problem of difficult-weaning patients with Non neurogenic disease in ICU. | From June 1st 2017 to June 30 2020
  Based on nutritional support, Cardiopulmonary rehabilitation and Levosimendan Bundle measures, and making beside checklist of patients with difficult ventilator weaning; Implementation of nutritional risk, respiratory function, and cardiac function assessment prior to weaning; Regulate the procedure to solve the problem of difficult-weaning patients with Non neurogenic disease in ICU. Thereby,improve the success rate of weaning patients, so as to shorten the ICU hospitalization time, reduce medical costs, reduce the complications of mechanical ventilation, improve the patient's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Xinke, Study Director — study principal investigator Shenzhen Second Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No